CLINICAL TRIAL: NCT06271642
Title: Impact of Vibrating Device Distraction on Mechanical Pain Thresholds Induced by Needle Sham
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 73822
Record Dates: First submitted 2024-02-06; First posted 2024-02-22 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Pain; Anxiety
Keywords: vibrating device
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bluetooth Haptic Device (Experimental Frequency) + Needle Sham (Experimental): Bluetooth Haptic Device with experimental vibrating frequency will be placed on the arm of the participant, with weighted pinpricks with fixed stimulus intensities will be applied.
  Interventions: Behavioral: Bluetooth Haptic Device (Experimental Frequency) + Needle Sham only
- Bluetooth Haptic Device (Control Frequency) + Needle Sham (Sham Comparator): Bluetooth Haptic Device with control vibrating frequency will be placed on the arm of the participant, with weighted pinpricks with fixed stimulus intensities will be applied.
  Interventions: Behavioral: Bluetooth Haptic Device (Control Frequency) + Needle Sham only

INTERVENTIONS:
Behavioral: Bluetooth Haptic Device (Experimental Frequency) + Needle Sham only — Participants will have the Bluetooth Haptic Device with experimental Frequency placed on their arm and randomized to a series of 4 different vibration patterns/frequencies. Mechanical pain threshold (MPT) will be measure using custom-made weighted pinprick stimuli as a set of five pinprick mechanical stimulators with fixed stimulus intensities (flat contact area of 0.2mm diameter) with forces of 32, 64, 128, 256, and 512mN. The stimulators will be applied at a rate of 2s on, 2s off in a randomized order on participants' forearms until the first sensation of pain is reached and will then be done in descending order until the sensation of pain disappears. This procedure will be repeated five times of ascending and descending stimuli served as pinprick pain threshold on 1 arm at 4 different frequencies/patterns in the BHD.
  Arms: Bluetooth Haptic Device (Experimental Frequency) + Needle Sham
Behavioral: Bluetooth Haptic Device (Control Frequency) + Needle Sham only — Participants will have the Bluetooth Haptic Device with control frequency placed on their arm. They will be randomized to a series of 4 different vibration patterns/frequencies. Mechanical pain threshold (MPT) will be measure using custom-made weighted pinprick stimuli as a set of five pinprick mechanical stimulators with fixed stimulus intensities (flat contact area of 0.2mm diameter) with forces of 32, 64, 128, 256, and 512mN. The stimulators will be applied at a rate of 2s on, 2s off in a randomized order on participants' forearms until the first sensation of pain is reached and will then be done in descending order until the sensation of pain disappears. This procedure will be repeated five times of ascending and descending stimuli served as pinprick pain threshold on 1 arm at 4 different frequencies/patterns in the BHD.
  Arms: Bluetooth Haptic Device (Control Frequency) + Needle Sham

SUMMARY:
This is a prospective, crossover study of healthy participants evaluating the mechanical pain threshold for weighted pinprick stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age
* English speaking
* Hearing intact

Exclusion Criteria:

* History of chronic pain or acute pain syndromes
* History of neurological, internal or psychiatric conditions
* Has active infections on arms and hand
* Has hearing loss
* Is pregnant
* Is currently taking beta blockers, chronotropic heart medications, or opioids or other prescription pain medications

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2024-06-06 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
Mechanical Pain Threshold | immediately after intervention
  Mechanical Pain Threshold will be measured using custom-made weighted pinprick stimuli as a set of seven pinprick mechanical stimulators with fixed stimulus intensities (flat contact area of 0.2mm diameter) with forces of 8, 16, 32, 64, 128, 256, and 512mN.

SECONDARY OUTCOMES:
Mechanical pain sensitivity | immediately after intervention
  Mechanical pain sensitivity will be taken immediately following each group of levels tests from 0-10; 0=no pain to 10=worst pain ever experienced.
Anxiety scores | immediately after intervention
  Anxiety level measured by a numerical rating scale (NRS) from 0-10. Scale ranges from 0-10, with higher scores indicating higher anxiety levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Lucile Parkard Children's Hospital, Stanford, California, United States